CLINICAL TRIAL: NCT07284810
Title: Tracking Reported Activities and Needs for Self-care, Function, Outcomes, Relief, and Mood
Brief Title: Tracking Self-Reported Functional Needs and Quality of Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Webster, Clinical Operations Manager, Cionic, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIONIC-07-001
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Upper Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cionic Neural Sleeve NS-200 (Experimental): Participants will wear the device and receive stimulation assistance during the exercise and walking sessions.
  Interventions: Device: Cionic Neural Sleeve System

INTERVENTIONS:
Device: Cionic Neural Sleeve System — The sleeve assists participants during physical activity by delivering electrical stimulation that helps contract the necessary muscles at the correct time to improve movement.

SUMMARY:
The study aims to characterize the population of Cionic Neural Sleeve users and assess their health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the United States
* New customer awaiting the Cionic Neural Sleeve

Exclusion Criteria:

* Implanted demand-type cardiac pacemaker or defibrillator
* Malignant tumor or existing thrombosis in the impacted or more impacted leg
* Fracture or dislocation in the impacted or more impacted leg that could be adversely affected by motion from stimulation

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | Day 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12
  Health related quality of life will be assessed by the EuroQol-5 Dimensions 5-Levels (EQ-5D-5L), a 6-item instrument to describe health in 5 dimensions. Each response of the EQ-5D-5L is assigned a numerical value from 1 to 5, with 1 being "no problems" and 5 being "extreme problems".

OTHER OUTCOMES:
Wear time | Every month from enrollment to the end of study at 12 months
  Wear time measured by the usage log of the device, measured in hours.
Device adherence | Every month from enrollment to the end of study at 12 months
  Wear time measured by the usage log of the device, measured in step count.
Spasticity | Day 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12
  The impact of spasticity on walking or movement will be collected. The score ranges from 0 - 5, with a higher score reflecting more severe spasticity.
Urinary Incontinence | Day 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12
  The frequency of urinary leaking will be collected. The score ranges from 1 - 5, with a higher score reflecting more frequent urinary incontinence.
Fatigue | Day 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12
  The impact of fatigue will be collected. The score ranges from 1 - 5, with a higher score reflecting more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- CIONIC, San Francisco, California, United States